CLINICAL TRIAL: NCT00160589
Title: A Multicentre, Double-blind, Parallel, Randomized, Placebo-controlled Study : Evaluation of the Efficacy and Safety of Levocetirizine 5 mg and Desloratadine 5 mg Administered Orally as Capsules Once Daily, in the Morning, Over 2 Weeks in Patients Suffering From Allergic Rhinitis (AR)
Brief Title: LEADER (LEvocetirizine And DEsloratadine in Allergic Rhinitis)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A00401; EudraCT2004-002823-42; LEADER
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Allergic Rhinits, Symptoms (sneezing, rhinorrhea, nasal/ocular pruritus, nasal congestion), LEADER, Xyzal, Levocetirizine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Sneezing; Rhinorrhea; Nasal Obstruction | interventions — levocetirizine

INTERVENTIONS:
Drug: Levocetirizine

SUMMARY:
Two weeks study to evaluate the efficacy and safety of Levocetirizine and Desloratadine in patients suffering from Allergic Rhinitis (AR)

ELIGIBILITY:
Inclusion Criteria:

* At least 2-year history of Allergic Rhinitis that became symptomatic during the annual grass pollen season.
* A skin test for grass pollens positive:
* Have rhinitis symptoms of such severity that the mean T4SS over the baseline period must be 6.

Exclusion Criteria:

* Have an associated asthma requiring corticosteroid treatment,
* Have an atopic dermatitis or an urticaria requiring an antihistamine treatment or the administration of oral or topical corticosteroids,

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 729
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline of T4SS (four symptoms score) over two weeks of treatment

SECONDARY OUTCOMES:
Clinical efficacy over the first and over two weeks of treatment measured by symptoms (scored and individuals); Onset of action; Safety

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma